CLINICAL TRIAL: NCT00077168
Title: Randomised Trial Testing Observation (No Radiotherapy) Against Radiotherapy In Women With Low-Risk Completely Excised ER Positive Ductal Carcinoma In Situ (DCIS) Of The Breast On Adjuvant Endocrine Therapy
Brief Title: Adjuvant Radiation Therapy Compared With Observation After Surgery in Treating Women With Estrogen Receptor Positive or Progesterone Receptor Positive Ductal Carcinoma In Situ of the Breast Who Are Receiving Tamoxifen or Anastrozole
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000349580; ICR-DCIS-II; EU-20341
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Anastrozole; Tamoxifen; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: anastrozole
Drug: tamoxifen citrate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether radiation therapy after surgery is effective in preventing a recurrence of ductal carcinoma in situ.

PURPOSE: This randomized phase II trial is studying adjuvant radiation therapy to see how well it works compared to observation after surgery in treating women with estrogen receptor positive or progesterone receptor positive ductal carcinoma in situ and are also receiving either tamoxifen or anastrozole.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare ipsilateral tumor relapse and breast cancer metastases in women with completely excised low-risk estrogen receptor- or progesterone receptor-positive ductal carcinoma in situ of the breast receiving adjuvant tamoxifen or anastrozole and treated with adjuvant radiotherapy vs observation alone.
* Compare the quality of life of patients treated with these regimens.

Secondary

* Determine the minimal surgical margins required to minimize the local recurrence rate in patients treated with these regimens.
* Identify molecular markers that predict ipsilateral tumor recurrence in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

All patients receive adjuvant tamoxifen or anastrozole for 5 years.

* Arm I: Patients undergo radiotherapy 5 days a week for 3 or 5 weeks.
* Arm II: Patients undergo observation alone. Quality of life is assessed at baseline, at 6 months, and then at 1, 2, and 5 years.

Patients are followed every 6 months for 1 year and then annually for up to 10 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 2,000 patients (1,000 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of unifocal ductal carcinoma in situ of the breast without an invasive component

  * Microinvasion (defined as 1 or more foci of invasion each < 1 mm) allowed
* Prior complete microscopic excision (within the past 6 months) with a minimum radial margin of 1 mm by specimen x-ray required
* Maximum microscopic tumor diameter < 30 mm (< 15 mm if grade 3 tumor)
* Planning to receive adjuvant tamoxifen or anastrozole for 5 years

  * Eligible patients may receive adjuvant endocrine therapy on ICR-IBIS-II
* Hormone receptor status:

  * Estrogen receptor positive OR
  * Progesterone receptor positive
  * More than 10% tumor staining for receptor OR a cutpoint of ≥ 2

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Premenopausal, perimenopausal, or postmenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No prior deep vein thrombosis

Pulmonary

* No prior pulmonary embolus

Other

* No unexplained postmenopausal bleeding
* No contraindication to full-dose radiotherapy to the breast
* No other cancer within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics
* No prior tamoxifen or raloxifene use for more than 3 months in duration

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior mastectomy

Other

* No concurrent anticoagulants

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2004-04; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Local tumor control (invasive and in situ local recurrence)

SECONDARY OUTCOMES:
Mastectomy rate
Pattern of relapse in the breast
Contralateral primary
Breast cancer metastases
Mortality
Quality of life
Molecular markers that predict ipsilateral tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Kaggwa — Institute of Cancer Research, United Kingdom
Locations (29):
- United Kingdom (29):
  - Frenchay Hospital at North Bristol NHS Trust, Bristol, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Broomfield Hospital, Broomefield, England
  - Chelmsford and Essex Centre, Chelmsford, England
  - Essex County Hospital, Colchester, England
  - Derbyshire Royal Infirmary, Derby, England
  - Queen's Hospital, Derby, England
  - Dorset County Hospital, Dorchester, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Lincoln County Hospital, Lincoln, England
  - Charing Cross Hospital, London, England
  - South Manchester University Hospital, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Derriford Hospital, Plymouth, England
  - Poole Hospital NHS Trust, Poole Dorset, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Scarborough General Hospital, Scarborough, England
  - University Hospital of North Tees, Stockton-on-Tees, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Torbay Hospital, Torquay Devon, England
  - Hillingdon Hospital, Uxbridge, England
  - Worcester Royal Hospital, Worcester, England
  - Aberdeen Royal Infirmary at NHS Grampian, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - University of Glasgow, Glasgow, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - University Hospital of Wales, Cardiff, Wales